CLINICAL TRIAL: NCT00396292
Title: Comparison of the Safety and Efficacy of Intravenous Iron vs Oral Iron in Subjects Who Display Postpartum Anemia
Brief Title: Comparison of the Safety and Efficacy of Intravenous Iron Versus Oral Iron in Subjects Who Display Postpartum Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VIT03001
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Results first posted 2013-12-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Anemia
Keywords: Anemia; postpartum; Postpartum anemia
MeSH Terms: conditions — Anemia | interventions — Iron; ferrous sulfate; ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIT-45 (Experimental): A maximum of 1,000 mg iron as IV VIT-45 given at weekly intervals until the the cumulative dose has been reached or a maximum of 2,500 mg has been administered
  Interventions: Drug: VIT-45
- Oral iron tablets (Active Comparator): 325 mg tablets (65 mg elemental iron) with instructions to take 1 tablet by mouth (PO) TID with 8 ounces of tap water, 1 hour before meals from Day 0 until Day 42
  Interventions: Drug: Oral iron tablets

INTERVENTIONS:
Drug: Oral iron tablets — 325 mg tablets (65 mg elemental iron) with instructions to take 1 tablet by mouth (PO) TID with 8 ounces of tap water, 1 hour before meals from Day 0 until Day 42
  Other Names: Ferrous Sulfate
  Arms: Oral iron tablets
Drug: VIT-45 — A maximum of 1,000 mg iron as IV VIT-45 given at weekly intervals until the the cumulative dose has been reached or a maximum of 2,500 mg has been administered
  Arms: VIT-45

SUMMARY:
This study compares the safety and efficacy of intravenous iron vs oral iron in subjects who display postpartum anemia.

DETAILED DESCRIPTION:
This is an open label, Phase III, randomized, active controlled study of intravenous iron vs oral iron in anemic post partum patients.

ELIGIBILITY:
Inclusion Criteria:

* Female Subjects able to give consent
* Post partum patients
* Baseline Hbg< /= 10
* Agree to practice birth control
* Demonstrate willingness to comply with protocol restrictions

Exclusion Criteria:

* Known hypersensitivity reaction to oral or IV iron (VIT-45)
* Documented history of discontinuing oral iron
* Significant bleeding
* History of anemia other that iron deficiency anemia
* Severe Psychiatric disorders
* Active severe infection
* Known Hepatitis B antigen or Hep C viral antibody or active hepatitis
* Known HIV antibody
* Received investigational product within 30 days
* Alcohol abuse
* Hemochromatosis or other iron storage disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luitpold Pharmaceuticals, Norristown, Pennsylvania, United States

REFERENCES:
- [Result] Baker JB, Seid MH, Van Wyck DB, Mangione A. Ferric Carboxymaltose, a New IV Iron Agent for Postpartum Anemia. Society for the Advancement of Blood Management 6th Annual Meeting 2007.
- [Result] Baker JB, Seid MH, Van Wyck DB, Dinh Q. Ferric Carboxymaltose, a New IV Iron Agent for Treating Postpartum Women with Iron Deficiency Anemia. Society for the Advancement of Blood Management 6th Annual Meeting 2007.
- [Derived] Van Wyck DB, Martens MG, Seid MH, Baker JB, Mangione A. Intravenous ferric carboxymaltose compared with oral iron in the treatment of postpartum anemia: a randomized controlled trial. Obstet Gynecol. 2007 Aug;110(2 Pt 1):267-78. doi: 10.1097/01.AOG.0000275286.03283.18. PMID 17666600

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitals and medical clinics
Pre-assignment Details: 8 subjects randomized to VIT-45 were discontinued prior to dosing due to subject request (3 subjects), lost to follow-up (2 subjects), 'other reasons' (2 subjects), and physician decision (1 subject). The 1 subject that was randomized to oral iron was lost to follow-up.
Period: Overall Study
Arm/Group | VIT-45 | Oral Iron Tablets
Started | 174 | 178
Completed | 165 | 162
Not Completed | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIT-45 | Oral Iron Tablets | Total
Number analyzed (Participants) | 174 | 178 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 159 | 162 | 321
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.93 (6.36) | 26.03 (5.95) | 26.41 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 178 | 352
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 174 | 178 | 352

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved 'Success' Meaning a ≥ 2.0 Increase in Hemoglobin
Time Frame: anytime between baseline and the end of study or time to intervention
Population: Modified Intent to Treat Population defined as subjects who received at least 1 dose of randomized study medication, had at least 1 post-baseline hemoglobin assessment, and had postpartum anemia characterized by an average of the 2 baseline central laboratory hemoglobin being <11.0 g/dL
Measure: Number; unit: participants
Arm/Group | VIT-45 | Oral Iron Tablets
Number analyzed (Participants) | 168 | 169
participants | 162 | 159

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | VIT-45 | Oral Iron Tablets
Serious Adverse Events (participants affected / at risk) | 4/174 | 4/178
Other Adverse Events (participants affected / at risk) | 40/174 | 61/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VIT-45 (N=174) | Oral Iron Tablets (N=178)
Peripartum cardiomyopathy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Postoperative infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VIT-45 (N=174) | Oral Iron Tablets (N=178)
Constipation (Gastrointestinal disorders) | 7 | 25
Nausea (Gastrointestinal disorders) | 3 | 15
Headache (Nervous system disorders) | 30 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less